CLINICAL TRIAL: NCT00314652
Title: A Double-Blind Placebo-Controlled Study of Buprenorphine Transdermal System (BTDS) in Patients With Osteoarthritis of the Hip or Knee
Brief Title: Safety and Efficacy of the Buprenorphine Transdermal Delivery System in Subjects With Osteoarthritis Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP99-0203
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; chronic pain; opioid; transdermal
MeSH Terms: conditions — Osteoarthritis; Chronic Pain

INTERVENTIONS:
Drug: Buprenorphine transdermal delivery system

SUMMARY:
The objective of this study is to assess the safety and efficacy of the buprenorphine transdermal system (5, 10, and 20 mg) in comparison to placebo transdermal system in subjects with osteoarthritis pain. The double-blind treatment intervention duration is 28 days.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over twenty-five years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain. Transdermal systems may offer advantages over currently indicated oral products including ease and convenience of use, improved compliance, possible reduction in patient care, and prolonged and consistent delivery of drug.

ELIGIBILITY:
Inclusion Criteria:

* documented history and/or radiologic evidence of chronic osteoarthritis of the hip or knee.
* receiving opioid therapy for osteoarthritis-related pain within the past year or have experienced pain that was inadequately controlled with a full standard dose of NSAIDs.

Exclusion Criteria:

* receiving opioids at an average daily dose of greater than 90 mg of oral morphine equivalents or patients receiving more than 12 tablets or capsules per day of short-acting opioid-containing products
* scheduled to have surgery (including dental) during the study period that involved the use of pre- and/or postoperative analgesics or anesthetics.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 1999-06; Study Completion 1999-10

PRIMARY OUTCOMES:
Percentage of patients who were treated successfully for pain management
a patient fails if he or she discontinues early due to ineffective treatment or has a Patient Satisfaction Scale score of poor or fair at the final visit

SECONDARY OUTCOMES:
Average pain intensity and patient satisfaction scores
Incidence of early discontinuation due to lack of efficacy
Time to early discontinuation due to lack of efficacy
Dose level at end of titration
Investigator's assessment of therapeutic response
Diary pain scores

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Hawthorne & York, International, Ltd., Phoenix, Arizona
  - Arizona Research Center, LLC, Phoenix, Arizona
  - ACRC/Arizona Clinical Research, Tucson, Arizona
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - San Diego Arthritis and Osteoporosis Research, San Diego, California
  - Scripps Clinic Rancho Bernardo, San Diego, California
  - Clinical Research Consultants, Inc., Trumbull, Connecticut
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - University Clinical Research, DeLand, Florida
  - Gainesville Clinical Research Center, Gainesville, Florida
  - Physicians Research Associates Jacksonville, Jacksonville, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Gold Coast Research, Inc., Weston, Florida
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Westside Family Medical Center, Kalamazoo, Michigan
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - NJP Clinical Research, Passaic, New Jersey
  - PW Clinical Research, LLC, Winston-Salem, North Carolina
  - New Century Research Center, Ltd., Beaverbrook, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Mid-South Clinical Research Institute, Memphis, Tennessee
  - Advanced Clinical Research, Salt Lake City, Utah